CLINICAL TRIAL: NCT02561975
Title: Adaptation of Alveolar-capillary Diffusion at Effort of Subjects Suffering From Complex Congenital Heart Disease
Acronym: CAR-DIFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9375
Record Dates: First submitted 2015-01-12; First posted 2015-09-29 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Complex Congenital Heart Disease; Single Ventricle With Fontan Circulation or Bicavo-bipulmonary Bypass; Systemic Right Ventricle; Pulmonary Failure
Keywords: Double pulmonary diffusing capacity to carbon monoxyd (CO) associated to nitric oxide (NO); Evolution of membrane and capillar damages; Early pronostic value of congenital heart disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient suffering from complex congenital heart disease (Experimental)
  Interventions: Other: Double pulmonary diffusing

INTERVENTIONS:
Other: Double pulmonary diffusing — Measure of double pulmonary diffusing will be done as the single-breath test: the patient will be seated and connected to device by an oral tip. Measure begins by a maximal inhalation of a gas mixture (0.28% of CO, 14% of He, 21% of O2,450 ppm of NO/N2 and 40ppm of NO).After, the patient will maintain an apnea of 4 secondes and will breathe out in oral tip until his residual capacity.
  With the expired air, some parameters will be assessed:
  * Alveolar volume (VA)
  * Membrane ductance (Dm) and pulmonar capillary volume (values adjusted by Haemoglobin)
  * Values of TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO et Dm/Vc

SUMMARY:
An injury of haematosis in post ischemic chronic heart failure limits the clinic tolerance.

There is a correlation between injury of pulmonary diffusing, chronic heart failure intensity and aerobic physic ability evaluated by an heart-rate maximal exercise tolerance test (VO2 max). This injury is a new follow-up parameter of cardiac function for the adult.

The nature of damage (vascular or membrane) can be determined by the measure of double pulmonary diffusing capacity to carbon monoxide (CO) associated to nitric oxide (NO).

Today, in chronic heart failure consecutive to a congenital heart disease, there is no data on evolution of membrane and capillar factors.It is impossible to predict if membrane damage will be the best factor correlated to the VO2max in patients suffering from complex congenital heart disease.

Assessing these parameters could be an comparative evaluation of heart-rate exercise tolerance test with VO2max and an early control of his damage without risks related to heart-rate maximal exercise and independently of age, sex, hemoglobin, type of heart disease.These results would have an early prognostic value that would permit to refine the follow-up and the treatment.

The main objective of this trial is to assess the statistic correlation between the membrane injury of alveolar-capillary diffusing at rest and aerobic physic ability restriction in children and adults suffering from complex congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 8 years- female and male patients
* Heart-rate exercise tolerance test planned in the usual patient's follow-up
* Congenital heart disease: single ventricle with Fontan circulation or bicavo-bipulmonary bypass or systemic right ventricle or pulmonary failure

Exclusion Criteria:

* Chronic or acute intercurrent respiratory disease
* In exclusion period in relation with another trial or for
* Participation to another study
* Patient doesn't benefit from an insurance disease regimen
* Pregnant woman or breast-feeding, law-protected person, vulnerable person

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Membrane ductance (Dm) correlated with VO2max | at the time of evaluation at rest (15 minutes before exercise)
  membrane ductance (Dm) is assessed by double pulmonary diffusing at rest

SECONDARY OUTCOMES:
capillary pulmonary recruitment during exercise correlated with VO2max. (capillary pulmonary volume 3 minutes after the end of a maximal exercise minus capillary pulmonary volume at rest) | at the time of evaluation at rest (15 minutes before exercise) and 3 minutes after the end of a maximal exercise
  capillary pulmonary volume 3 minutes after the end of a maximal exercise minus capillary pulmonary volume at rest
parameters assessed during measure TLCO/TLNO of double pulmonary diffusing at rest correlated with electrocardiographic parameters | at the time of evaluation at rest (15 minutes before exercise)
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO and Dm/Vc
parameters assessed during measure TLCO/TLNO of double pulmonary diffusing 3 minutes after the end of a maximal exercise correlated with electrocardiographic parameters | 3 minutes after the end of a maximal exercise
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO et Dm/Vc
parameters assessed during measure TLCO/TLNO of double pulmonary diffusing 10 minutes after the end of a maximal exercise correlated with electrocardiographic parameters | 10 minutes after the end of a maximal exercise
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO et Dm/Vc
parameters assessed during measure TLCO/TLNO of double pulmonary diffusing at rest correlated with VO2max | at the time of evaluation at rest (15 minutes before exercise)
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO and Dm/Vc
parameters assessed during measure TLCO/TLNO of double pulmonary diffusing at rest correlated with clinic dyspnea (NYHA) | at the time of evaluation at rest (15 minutes before exercise)
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO and Dm/Vc
parameters assessed during measure TLCO/TLNO of double pulmonary diffusing 3 minutes after the end of a maximal exercise correlated with VO2max | 3 minutes after the end of a maximal exercise
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO et Dm/Vc
diffusing 3 minutes after the end of a maximal exercise correlated with clinic dyspnea (NYHA) | 3 minutes after the end of a maximal exercise
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO et Dm/Vc
parameters assessed during measure TLCO/TLNO of double pulmonary diffusing 10 minutes after the end of a maximal exercise correlated with VO2max | 10 minutes after the end of a maximal exercise
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO et Dm/Vc
diffusing 10 minutes after the end of a maximal exercise correlated with clinic dyspnea (NYHA) | 10 minutes after the end of a maximal exercise
  parameters assessed during measure TLCO/TLNO of double diffusing are TLCO, TLCO/VA, TLNO, TLNO/VA Vc, Dm, Vc/VA, Dm/VA, TLNO/TLCO et Dm/Vc

CONTACTS AND LOCATIONS:
Overall Officials: Stephan MATECKI, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France